CLINICAL TRIAL: NCT02202005
Title: A Multiple Dose, Open Label, Pivotal, 4 Period, 2 Treatment, Sequence Full Replicative Crossover Study to Assess the Bioequivalence (BE) of TEVA's Generic Once Daily Nevirapine 400 mg Prolonged Release (PR) Formulation Compared With the Approved Reference Product Viramune® 400 mg Prolonged Release Tablets Under Fasted Conditions in HIV1 Infected Patients
Brief Title: Multiple Dose BE Study With Nevirapine 400mg PR Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ratiopharm GmbH (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: NEVIR5U14EU; 2014-002247-18 (EudraCT Number)
Record Dates: First submitted 2014-07-24; First posted 2014-07-28 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: HIV-1
Keywords: Bioequivalence
MeSH Terms: interventions — Nevirapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nevirapine (Experimental)
  Interventions: Drug: Nevirapine; Drug: Viramune®
- Viramune® (Active Comparator)
  Interventions: Drug: Nevirapine; Drug: Viramune®

INTERVENTIONS:
Drug: Nevirapine — Nevirapine 400mg PR tablet
Drug: Viramune® — Viramune® 400 mg Retardtabletten

SUMMARY:
The objective of this steady state pivotal study is to compare the rate and extent of absorption and to evaluate Bioequivalence of test drug compared to the approved reference product in HIV infected individuals

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated written informed consent prior to admission to the study
2. HIV1 infected males or females of 18 to 65 years, nonsmoker (use of cannabis may be accepted)
3. Body weight ≥ 50.0 kg and BMI ≥ 18.0 and ≤ 32.0 kg/m2
4. Absence of clinically significant history of neurological, endocrinal, cardiovascular, pulmonary, haematological, psychiatric, gastrointestinal, renal, hepatic, obstructive disorders, cholestasis, and metabolic disease
5. Treatment with a stable nevirapine based combination regimen for at least the preceding 12 weeks (or 6 weeks if switched from an antiretroviral regimen containing two nucleoside analogues and efavirenz)
6. Background HIV therapy with a stable antiretroviral regimen that is recommended in combination with nevirapine according to British HIV Association clinical guidelines:

   1. Abacavir and lamivudine {ABC/3TC} as fixed dose combination Kivexa
   2. Tenofovir and emtricitabine {TDF/FTC} Truvada
   3. Zidovudine and lamivudine {AZT/3TC} - Combivir, OR
   4. Tenofovir and lamivudine as separately prescribed components and kept constant (in combination and dosage) throughout the whole course of the study
7. An HIV viral load < 50 copies/mL in preceding 3 months and at screening
8. A CD4+ Tcell count > 50 cell/mm3
9. Acceptable screening laboratory values that indicate adequate baseline organ function
10. Willingness to abstain from ingesting medications that are listed as contraindicated for nevirapine during the whole course of the study
11. Capable of completing patient diaries
12. Capable and willing to come back for PK assessments and follow up
13. Willingness to refrain from excessive physical activity during the trial
14. Willingness of male study participants to not father a child during and throughout the study. To prevent a pregnancy of the female partner, both the male study participant and the female partner need to take appropriate contraceptives to prevent pregnancy during the study.

Exclusion Criteria:

1. Infection with HIV2 or HIV1 group O.
2. Current treatment with an HIV protease inhibitor
3. Participation in any other study within 30 days of Day 1, or intention to participate in another study during participation in this study.
4. Male and female patients who are not willing to use male or female condoms to prevent HIV transmission
5. Female patients of childbearing potential who:

   1. Have a positive serum pregnancy test at screening.
   2. Are breast feeding.
   3. Are planning to become pregnant
   4. Are not willing to take appropriate measures to prevent pregnancy during the study
6. Females who do not use an acceptable contraceptive regimen or confirm total abstinence will be allowed to participate in this study only if they are not considered to be of childbearing potential
7. Laboratory parameters > DAIDS grade 2 Coagulation
8. Laboratory parameters > DAIDS grade 2 Total triglycerides
9. Hypersensitivity to the active substance or any ingredients of the test or reference investigational products or chemically related compounds.
10. Contraindication to Nevirapine
11. Relevant history or current condition, illness that might interfere with drug absorption, distribution, metabolism or excretion
12. Use of concomitant medication (other than the stable background antiretroviral HIV therapy) that may interfere with the pharmacokinetics of nevirapine and/or the background antiretroviral HIV therapy)
13. Intake of products containing St. John's Wort from 14 days before treatment with study medication (Day 1) and not willing to abstain from it throughout the study until after the last study visit

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2014-08; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations by AUC0 τ,ss (area under the concentration time curve) | Days 14, 28, 42, 56
Cτ,ss (defined as concentration at the end of dosing interval) | Days 14, 28, 42, 56
Cmax,ss (maximum observed plasma concentration) | Days 14, 28, 42, 56

SECONDARY OUTCOMES:
Percentage of fluctuation over one dosing interval at steady state (Fl(%) | Days 14, 28, 42, 56
Tmax,ss (the time to maximum plasma concentration at steady state) | Days 14, 28, 42, 56
Cmin,ss (minimum plasma concentration at steady state) | Days 14, 28, 42, 56
Average plasma drug concentration | Days 14, 28, 42, 56

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Principal Investigator — Chelsea and Westminster NHS Foundation Trust
Locations (1):
- Chelsea and Westminster NHS Foundation Trust, London, United Kingdom